CLINICAL TRIAL: NCT06745219
Title: Herombopag for the Prevention of Radio-chemotherapy Induced Thrombocytopenia in Cervical Cancer: A Single-arm Phase II Clinical Trial
Brief Title: Herombopag for the Prevention of Radio-chemotherapy Induced Thrombocytopenia in Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, xiaofanli, MD., Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024YJZ53
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Thrombopenia; Cervical Cancer; Radiotherapy Side Effect; Chemotherapeutic Toxicity
MeSH Terms: conditions — Thrombocytopenia; Uterine Cervical Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Herombopag (Experimental): Cervical cancer patients who developed thrombopenia after receiving radiotherapy and platinum-based chemotherapy were enrolled
  Interventions: Drug: herombopag

INTERVENTIONS:
Drug: herombopag — receive harombopag for the prevention of thrombocytopenia in the next cycle of chemotherapy
  Other Names: Platelet receptor agonists

SUMMARY:
Exploring and evaluating the efficacy of herombopag in preventing thrombocytopenia due to radiotherapy for cervical cancer

DETAILED DESCRIPTION:
Thrombocytopenia is a relatively common adverse effect for cancer treatment. At present, for the secondary prevention of thrombocytopenia associated with tumor therapy, TPO-RA drugs have been included in the Level III recommendation of the "Thrombocytopenia Diagnosis and Treatment Guidelines for Cancer Treatment (2022 Edition)".

Herombopag, a new generation of thrombopoietin receptor agonist, is a Class 1 innovative drug independently developed in China, which has been approved in June 2021 for the indication of chronic primary immune thrombocytopenia with poor response to previous treatments of glucocorticoids and immunoglobulins, as well as severe aplastic anemia with poor efficacy of immunosuppressive treatments. As an oral medication, this drug is more convenient and safer than traditional injectable preparations. However, this drug has not been formally approved for the treatment of therapy-related thrombocytopenia.

This study is planned to enroll cervical cancer patients with thrombocytopenia due to radiotherapy combined with a three-week regimen of chemotherapy, and to evaluate the efficacy of herombopag in preventing thrombocytopenia in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the trial and sign the informed consent
2. Pathologically or cytologically confirmed cervical cancer
3. aged 18 years or older
4. ECOG performance score 0-1
5. Stage IB3-IVA according to 2018 FIGO stage
6. Patients receiving cisplatin-contained two-drug every-three week chemotherapy; minimum PLT value of the last chemotherapy <50×109/L, or ≥50 ×109/L, but <75×109/L, meeting at least one high risk factor for bleeding: previous bleeding history; receiving cisplatin, gemcitabine, cytarabiine, anthracycline chemotherapy; combination of targeting or chemotherapy drugs likely to cause thrombocytopenia; tumor bone marrow infiltration; receiving radiotherapy, such as long bone or flat bone (pelvic or sternum)
7. Survival expected to be ≥12 weeks, and can be treated with the concurrent chemotherapy regimen for at least one cycle
8. Participants of reproductive age who agree to use reliable contraceptive methods throughout the study period (including male or female condoms, contraceptive foam, contraceptive gel, contraceptive film, contraceptive paste, contraceptive suppository, abstinence from sex, and insertion of an IUD); Female subjects who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation or more than 1 year postmenopausal and male subjects who have undergone bilateral vasectomy or ligation are excluded
9. Participants can be treated with thrombopoietic drugs determined by researchers

Exclusion Criteria:

1. Participants with other diseases of hematopoietic system, including but not limited to leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma, and myelodysplastic syndrome
2. Participants with thrombocytopenia occurred within the last 6 months due to causes other than CTIT, including but not limited to chronic liver disease, hypersplenism, infection
3. Bone marrow invasion or metastasis
4. History of severe cardiovascular disease within the last 6 months, such as congestive heart failure (NYHA heart function score III-IV), arrhythmias known to increase the risk of thromboembolism such as atrial fibrillation, after coronary stenting, angioplasty, and para-coronary transplantation, etc
5. History of any arterial or venous thrombosis within the last 6 months
6. Severe bleeding within 2 weeks, such as gastrointestinal or central nervous system bleeding, vaginal bleeding, etc
7. Neutrophil absolute value <1.5×109/L, hemoglobin <80g/L, PLT<90× 109/L
8. Significantly abnormal liver function :TBIL>1.5ULN(upper limit of normal), >3ULN for patients known to have Gilbert syndrome; ALT>2.5ULN or AST>2.5ULN
9. Abnormal renal function: serum creatinine ≥1.5ULN or eGFR≤60 ml/min(Cockcroft-Gault formula)
10. Had received platelet infusion within 3 days
11. known or expected allergy or intolerance to the active ingredient or excipient of hetropopar ethanolamine tablets
12. HIV infected
13. Pregnant or lactating women
14. Participated in clinical trials of any other investigational drug or device within 28 days
15. Inability to swallow, inflammatory bowel disease, or uncontrollable nausea, vomiting, diarrhea, or other gastrointestinal disorders that severely affect the administration and absorption of medications
16. With a high risk for participants' safety or other conditions that may affect the efficacy evaluated by investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with PLT <75×109/L after the use of herombopag | Blood routine tests were conducted every three days within 14 days after the first day of chemotherapy
  number of participants with PLT <75×109/L/ all participants

SECONDARY OUTCOMES:
minimum value of platelet after chemotherapy | Blood routine tests were conducted every three days within 14 days after the first day of chemotherapy
  minimum value of platelet of every participants after chemotherapy for every participants
Change from baseline in PLT count minimum value | Blood routine tests were conducted every three days within 14 days after the first day of chemotherapy
  absolute value change from the maximum or minimum of platelet to baseline for every participants
Median duration of PLT <75×109/L | Blood routine tests were conducted every three days within 14 days after the first day of chemotherapy
  the days during the PLT <75×109/L of every participants
Median time to recovery of PLT to ≥100×109/L | Blood routine tests were conducted every three days within 14 days after the first day of chemotherapy
  the days during the PLT >100×109/L of every participants
Platelet count one day before the next chemotherapy | Blood routine tests were conducted every three days within 14 days after the first day of chemotherapy
  Platelet count one day before the next chemotherapy of every participants
Incidence of reduced intensity of next cycle chemotherapy due to decreased PLT | Blood routine tests were conducted every three days within 14 days after the first day of chemotherapy
  number of reduced intensity/number of no reduced intensity for next cycle chemotherapy due to decreased PLT

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Li, Dr, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu Y, Aravind S, Ranganathan G, Martin A, Nalysnyk L. Anemia and thrombocytopenia in patients undergoing chemotherapy for solid tumors: a descriptive study of a large outpatient oncology practice database, 2000-2007. Clin Ther. 2009;31 Pt 2:2416-32. doi: 10.1016/j.clinthera.2009.11.020. PMID 20110050
- [Result] Krigel RL, Palackdharry CS, Padavic K, Haas N, Kilpatrick D, Langer C, Comis R. Ifosfamide, carboplatin, and etoposide plus granulocyte-macrophage colony-stimulating factor: a phase I study with apparent activity in non-small-cell lung cancer. J Clin Oncol. 1994 Jun;12(6):1251-8. doi: 10.1200/JCO.1994.12.6.1251. PMID 8201386
- [Result] Veldhuis GJ, Willemse PH, Beijnen JH, Boonstra H, Piersma H, van der Graaf WT, de Vries EG. Paclitaxel, ifosfamide and cisplatin with granulocyte colony-stimulating factor or recombinant human interleukin 3 and granulocyte colony-stimulating factor in ovarian cancer: a feasibility study. Br J Cancer. 1997;75(5):703-9. doi: 10.1038/bjc.1997.125. PMID 9043028
- [Result] Elias A, Ryan L, Aisner J, Antman KH. Mesna, doxorubicin, ifosfamide, dacarbazine (MAID) regimen for adults with advanced sarcoma. Semin Oncol. 1990 Apr;17(2 Suppl 4):41-9. PMID 2110385
- [Result] Kim G, Ison G, McKee AE, Zhang H, Tang S, Gwise T, Sridhara R, Lee E, Tzou A, Philip R, Chiu HJ, Ricks TK, Palmby T, Russell AM, Ladouceur G, Pfuma E, Li H, Zhao L, Liu Q, Venugopal R, Ibrahim A, Pazdur R. FDA Approval Summary: Olaparib Monotherapy in Patients with Deleterious Germline BRCA-Mutated Advanced Ovarian Cancer Treated with Three or More Lines of Chemotherapy. Clin Cancer Res. 2015 Oct 1;21(19):4257-61. doi: 10.1158/1078-0432.CCR-15-0887. Epub 2015 Jul 17. PMID 26187614
- [Result] Mkhitaryan S, Danielyan S, Sargsyan L, Hakobyan L, Iskanyan S, Bardakchyan S, Papyan R, Arakelyan J, Sahakyan K, Avagyan T, Tananyan A, Muradyan A, Tamamyan G. Younger age and previous exposure to radiation therapy are correlated with the severity of chemotherapy-induced thrombocytopenia. Ecancermedicalscience. 2019 Feb 26;13:906. doi: 10.3332/ecancer.2019.906. eCollection 2019. PMID 30915164
- [Result] Penniment MG, De Ieso PB, Harvey JA, Stephens S, Au HJ, O'Callaghan CJ, Kneebone A, Ngan SY, Ward IG, Roy R, Smith JG, Nijjar T, Biagi JJ, Mulroy LA, Wong R; TROG 03.01/CCTG ES.2 group. Palliative chemoradiotherapy versus radiotherapy alone for dysphagia in advanced oesophageal cancer: a multicentre randomised controlled trial (TROG 03.01). Lancet Gastroenterol Hepatol. 2018 Feb;3(2):114-124. doi: 10.1016/S2468-1253(17)30363-1. Epub 2017 Dec 14. PMID 29248399
- [Result] Weycker D, Hatfield M, Grossman A, Hanau A, Lonshteyn A, Sharma A, Chandler D. Risk and consequences of chemotherapy-induced thrombocytopenia in US clinical practice. BMC Cancer. 2019 Feb 14;19(1):151. doi: 10.1186/s12885-019-5354-5. PMID 30764783
- [Result] Denduluri N, Lyman GH, Wang Y, Morrow PK, Barron R, Patt D, Bhowmik D, Li X, Bhor M, Fox P, Dhanda R, Saravanan S, Jiao X, Garcia J, Crawford J. Chemotherapy Dose Intensity and Overall Survival Among Patients With Advanced Breast or Ovarian Cancer. Clin Breast Cancer. 2018 Oct;18(5):380-386. doi: 10.1016/j.clbc.2018.02.003. Epub 2018 Feb 16. PMID 29622384
- [Result] Gernsheimer T. Chronic idiopathic thrombocytopenic purpura: mechanisms of pathogenesis. Oncologist. 2009 Jan;14(1):12-21. doi: 10.1634/theoncologist.2008-0132. Epub 2009 Jan 14. PMID 19144680
- [Result] Xie C, Zhao H, Bao X, Fu H, Lou L. Pharmacological characterization of hetrombopag, a novel orally active human thrombopoietin receptor agonist. J Cell Mol Med. 2018 Nov;22(11):5367-5377. doi: 10.1111/jcmm.13809. Epub 2018 Aug 29. PMID 30156363
- [Result] Mei H, Liu X, Li Y, Zhou H, Feng Y, Gao G, Cheng P, Huang R, Yang L, Hu J, Hou M, Yao Y, Liu L, Wang Y, Wu D, Zhang L, Zheng C, Shen X, Hu Q, Liu J, Jin J, Luo J, Zeng Y, Gao S, Zhang X, Zhou X, Shi Q, Xia R, Xie X, Jiang Z, Gao L, Bai Y, Li Y, Xiong J, Li R, Zou J, Niu T, Yang R, Hu Y. A multicenter, randomized phase III trial of hetrombopag: a novel thrombopoietin receptor agonist for the treatment of immune thrombocytopenia. J Hematol Oncol. 2021 Feb 25;14(1):37. doi: 10.1186/s13045-021-01047-9. PMID 33632264